CLINICAL TRIAL: NCT00004014
Title: Liposome-Encapsulated Doxorubicin (LED) in Hormone Refractory Prostate Carcinoma, Phase II
Brief Title: Liposomal Doxorubicin in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Cindy Connell, MD, PhD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO1898; P30CA043703 (NIH); CWRU-NEO-1898; NEOPHARM-LED-P2; NCI-G99-1558
Record Dates: First submitted 1999-11-01; First posted 2004-09-14 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride — Doxorubicin HCl liposome IV over 45 minutes every 3 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline and then every 9 weeks thereafter.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of liposomal doxorubicin in treating patients with prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the objective response rate of patients with hormone refractory prostate cancer treated with doxorubicin HCl liposome. II. Determine the toxic effects (including any cumulative cardiotoxicity) of this regimen in these patients. III. Assess the effect of this regimen on pain and quality of life of these patients.

OUTLINE: Patients receive doxorubicin HCl liposome IV over 45 minutes every 3 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline and then every 9 weeks thereafter. Patients are followed every 3 months.

PROJECTED ACCRUAL: Approximately 50 evaluable patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed hormone refractory prostate cancer Castrate serum testosterone levels less than 30 mg/dL occurring at least 4 weeks since prior flutamide or at least 6 weeks since prior bicalutamide Measurable or evaluable progressive disease Rising PSA involving two determinations (one at least 20 ng/mL if PSA is sole criterion) at least two weeks apart OR Increasing measurable or evaluable disease OR New metastasis

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL No hepatic insufficiency Renal: Creatinine no greater than 2.0 mg/dL No renal failure Cardiovascular: Cardiac ejection fraction at least 50% by radionuclide ventriculogram No myocardial infarction within the past year No active angina No congestive heart failure No arrhythmias requiring medication Other: No active peptic ulcers No uncontrolled infection or other serious medical condition that would prevent compliance with chemotherapy No uncontrolled diabetes No spinal cord compression or carcinomatous meningitis

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: No concurrent corticosteroid therapy Concurrent gonadotropin-releasing hormone analogue allowed Radiotherapy: At least 2 months since prior radiotherapy (not to a measurable lesion) Concurrent palliative radiotherapy allowed Surgery: Not specified

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 1999-04; Primary Completion 2000-01 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Effectiveness of liposomal doxorubicin in treating patients with prostate cancer that has not responded to hormone therapy. | Every 3 weeks, treatment continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline and then every 9 weeks thereafter. Patients are followed every 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Connell, MD, PhD, Study Chair — Ireland Cancer Center at University Hospitals/Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Cleveland, Ohio, United States